CLINICAL TRIAL: NCT05790694
Title: A Randomized, Double-blind, Placebo-controlled, Single-ascending-dose Phase I Clinical Study in Healthy Chinese Subjects to Evaluate the Safety, Tolerability and Pharmacokinetics of HBM9378 (SKB378) After Subcutaneous Administration.
Brief Title: A Trial of HBM9378 in Healthy Chinese Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harbour BioMed (Guangzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9378.1
Record Dates: First submitted 2023-02-27; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBM9378 (SKB378) Injection (Experimental): Dose: 20 mg/60 mg/200 mg/600 mg/900 mg Frequency: Once Injection subcutaneously
  Interventions: Drug: HBM9378 (SKB378) Injection
- Placebo (Placebo Comparator): Dose: 20 mg/60 mg/200 mg/600 mg/900 mg Frequency: Once Injection subcutaneously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HBM9378 (SKB378) Injection — Strength: 225 mg (1.5 mL)/vial
  Arms: HBM9378 (SKB378) Injection
Drug: Placebo — Strength: 225 mg (1.5 mL)/vial
  Arms: Placebo

SUMMARY:
The objective is to evaluate the safety, tolerability and pharmacokinetic profile of a single subcutaneous injection of HBM9378 (SKB378) at different doses in healthy Chinese subjects.

DETAILED DESCRIPTION:
The study will consist of one dose esclation part with a total of 5 dose levels. The Subjects will be randomized to receive HBM9378 as reflected by the guiding principle for the dose esclation/expansion phase. Each dose group includes a screening period, a baseline period, an observational period, and a safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained.
2. Healthy Chinese male and female subjects aged 18 to 50 years (both included) are enrolled, no clinically significant abnormalities.
3. Total body weight ≥45kg at screening, and body mass index(BMI)between 18 and 28 kg/m2 (inclusive).
4. Female subjects must meet one of the following criteria for participation in this study: Of non-childbearing potential ;
5. Male subjects and female subjects of childbearing potential must use an effective contraceptive method during their participation in this clinical study.
6. Can communicate successfully with the investigator and understand and comply with the requirements of this study.

Exclusion Criteria:

1. History of relevant allergy/hypersensitivity.
2. History of any of the following diseases:

   1. Any clinically significant comorbidity, as judged by the investigator.
   2. Clinical signs of active infection found at screening.
   3. Previous malignancy within the past 5 years.
   4. Acute or chronic bronchospastic disease within the past 3 years.
3. Subject who are currently suffering from any medical condition.
4. Subjects who have undergone organ transplantation.
5. Received immunosuppressive therapy within 6 months prior to randomization.
6. Received any biological product within 90 days or 5 half-lives (for other study drugs), whichever is longer, prior to randomization, or participated in another clinical study and received a study drug.
7. Received any drug within 4 weeks prior to randomization.
8. Subjects who had an immunization within 4 weeks prior to randomization; subjects who are scheduled to have an immunization during the study or within 4 weeks after the end of study.
9. Donated or lost 400 mL or more blood, or received transfusion of blood or any blood product within 60 days prior to randomization.
10. Subjects who are smokers or have used tobacco or nicotine-containing products within 3 months prior to randomization.
11. Subjects who regularly consumed alcohol within 3 months prior to screening, or who had consumed alcohol after screening and before administration.
12. Subjects who had been exposed to a tuberculosis (TB) patient within 6 months prior to randomization.
13. Subjects who had drug abuse or a positive urine drug screen within 12 months prior to randomization.
14. Pregnant or lactating women.
15. Positive hepatitis B surface antigen (HBsAg) or hepatitis C antibody test result, or clinically significantly abnormal syphilis serology test result.
16. History of immunodeficiency disease, including clinically significantly abnormal HIV antibody test result.
17. Clinically significantly abnormal vital signs, physical examination, chest radiography, electrocardiogram , or laboratory tests , as judged by the investigator.
18. In the investigator's judgment, may increase the risk to the subject.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-09-22 (Estimated); Study Completion 2023-09-22 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Strat of Treatment to end of study (approsimately 160days)
  Incidence and severity of adverse events
Pharmacokinetics-AUC0-last | Strat of Treatment to end of study (approsimately 160days)
  Area under the concentration-time curve from time 0 to last time point after HBM9378 administration
Pharmacokinetics-Tmax | Strat of Treatment to end of study (approsimately 160days)
  Time to Cmax of HBM9378
Pharmacokinetics-Cmax | Strat of Treatment to end of study (approsimately 160days)
  Maximum observed concentration of HBM9378
Pharmacokinetics-CL/F | Strat of Treatment to end of study (approsimately 160days)
  Apparent clearance of HBM9378
Pharmacokinetics-Vd/F | Strat of Treatment to end of study (approsimately 160days)
  Apparent volume of distribution during terminal phase of HBM9378
Pharmacokinetics-T1/2 | Strat of Treatment to end of study (approsimately 160days)
  Terminal elimination half-life of HBM9378

SECONDARY OUTCOMES:
Immunogenicity | Strat of Treatment to end of study (approsimately 160days)
  The percentage of patients with anti-drug antibodies after administration.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth People's Hospital of Chengdu, Sichuan, Chengdu, China